CLINICAL TRIAL: NCT07147244
Title: Guardians Receiving Information Through Navigators
Acronym: GRIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KDH Research & Communication (Industry)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025-02-04; 5R44MD016352-03 (NIH)
Record Dates: First submitted 2025-08-12; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Oral Health; Child; Adolescent; High-risk; Community Health Workers
Keywords: Community health workers; Adolescents; Oral Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment 1: Full GRIN course (Lessons 1-8) (Experimental): Lessons 1-8 of professional development training course for CHWs on dental health (GRIN)
  Interventions: Other: Treatment 1: Full GRIN course (Lessons 1-8)
- Treatment 2: Part 1 of GRIN (Lessons 1-4) (Experimental): Lessons 1-4 of professional development training course for CHWs on dental health (GRIN)
  Interventions: Other: Treatment 2: Part 1 of GRIN (Lessons 1-4)
- Treatment 3: Part 2 of GRIN (Lesson 1, 5-8) (Experimental): Lesson 1, 5-8 of professional development training course for CHWs on dental health (GRIN)
  Interventions: Other: Treatment 3: Part 2 of GRIN (Lesson 1, 5-8)
- Control 1 (No Intervention): No intervention
- Control 2 (No Intervention): No intervention
- Control 3 (No Intervention): No intervention

INTERVENTIONS:
Other: Treatment 1: Full GRIN course (Lessons 1-8) — multi module online training
  Arms: Treatment 1: Full GRIN course (Lessons 1-8)
Other: Treatment 2: Part 1 of GRIN (Lessons 1-4) — multi module online training
  Arms: Treatment 2: Part 1 of GRIN (Lessons 1-4)
Other: Treatment 3: Part 2 of GRIN (Lesson 1, 5-8) — multi module online training
  Arms: Treatment 3: Part 2 of GRIN (Lesson 1, 5-8)

SUMMARY:
A multi-arm study, experimental and control groups, to explore the impact of an online training program to help community health workers conduct effective outreach to support the dental health of high-risk youth via their guardians.

DETAILED DESCRIPTION:
The investigators will use a randomized, multi-group, pretest/posttest/follow-up design to test the efficacy of the Guardians Receiving Information Through Navigators (GRIN) course and explore the following research question: To what extent does exposure to the GRIN course relate to positive changes in community health workers' (CHWs') knowledge, attitudes and beliefs, perceived self-efficacy, and intent to conduct oral health care outreach to low-income Black guardians?

GRIN course will have eight full course lessons with text, video vignettes, and artificial intelligence (AI) avatar simulations. The study will consist of pretest, posttest, and 3-month follow-up surveys. CHWs assigned to the treatment group will be exposed to different doses of the intervention, including the full GRIN course (Lessons 1-8), Part 1 of GRIN (Lessons 1-4), or Part 2 of GRIN (Lesson1, 5-8). CHWs assigned to the control group will receive pages from the American Dental Association (ADA) website.

Researchers worked with subject matter experts, dental providers, and the intended audience to ensure the GRIN course reflects the specific needs of CHWs providing outreach to guardians of high-risk adolescents; minimize counter-productive duplications of services and resource expenditure; and create empowered opportunities for CHWs to improve their outreach skills.

The Principal Investigator (PI), with input from the subject matter experts and dental providers, developed necessary research materials, including the recruitment protocols, evaluation instrumentation, and human subjects consent materials . The PI also outlined the appropriate statistical analysis methods. All procedure documents will be reviewed by the KDH Research & Communication (KDHRC) Institutional Review Board before the evaluation launch.

Investigators will recruit participants through a multi-pronged recruitment strategy including 1) hiring a contractor to manage recruitment of CHWs by sharing study information and consent process to community-based organizations (CBOs) and other CHW organizations; 2) sharing the opportunity through the KDHRC CHW panel, which notifies subscribed CHWs about research opportunities; 3) recruiting at CHW conferences such as the National Association of Community Health Workers (NACHW) Annual Conference; and 4) posting on social media. Notifications and flyers will provide information about the goal of the study, participant eligibility, and a link to an eligibility form. Once a potential participant completes the eligibility form and s/he is eligible for the study, they will receive a link to a consent form located on a secure online platform.

The study will include up to 320 CHWs nationwide (160 treatment groups, 160 control groups). The recruitment contractor and sites will refer participants and may have access to potential participant information (e.g., name, email address) from their listservs, but will not have knowledge of who actually serves as study participants and will not have access to enrolled participants' data. KDHRC will remind participants that participation in the study is completely voluntary, that the referral sites will not have knowledge of who actually serves as study participants, and that his or her participation is no way tied to his or her position at and/or relationship with the site that shared referral materials with him or her.

Investigators will confirm consent for each participant and after confirming consent, will send participants the link to complete the pretest survey. Once the investigators receive the pretest survey, they will randomize each participant into the treatment group or control group using a 1:1 randomization. Investigators will alternate assigning each participant with completed pretest to the treatment groups or the control groups. Then, investigators will provide each treatment group participant with access to appropriate treatment link. The control group will be directed to ADA webpages. Participant responses to pretest and posttest survey measures will be linked using non-personal identifiers.

The investigators will download and export the data from Alchemer into encrypted Excel files and import the raw data into STATA. The investigators will match the pretest and posttest, and follow-up responses using the non-personal identifiers and conduct analyses to test for the effect of the GRIN course exposure on changes in CHWs' knowledge, attitudes and beliefs, perceived self-efficacy, and intent to conduct oral health care outreach to low-income guardians of high-risk adolescents.

The initial evaluation criterion is: Statistically significant (p<0.05) and positive relationship between exposure to GRIN course and increased knowledge among the intervention group in comparison to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years old.
* Must have six months of field experience. Investigators define "field experience" as conducting outreach activities in their community, for example, working with clients in a clinic, conducting home visits, or educating clients at health fairs or community events.
* Must be an active CHW/health educator/individual who conducts health outreach. Investigators define "active" as conducting outreach activities, such as working with clients in a clinic, conducting home visits, or educating clients at health fairs or community events, in the last six months.
* Must have Internet access either at home or at work (or at in-person session).

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge Pretest Score | Baseline
  We will ask participants multiple choice knowledge questions related to oral health which we will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 means a participant got zero questions correct while a score of 100 meant a participant got all questions correct. We will average these composite scores across all participants for both groups to create mean scores ranging from 0 to 100, the higher the score the more questions participants answered correctly.
Knowledge Posttest Score | Posttest (2 weeks after baseline)
  We will ask participants multiple choice knowledge questions related to oral health which we will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 means a participant got zero questions correct while a score of 100 means a participant got all questions correct. We will average these composite scores across all participants for both groups to create mean scores ranging from 0 to 100, the higher the score the more questions participants answered correctly.
Attitudes Pretest Score | Baseline
  We will ask all participants Likert-type scale questions about attitudes towards conducting oral health outreach. Each answer choice rating will range from 1 to 10, with higher ratings representing higher perceptions of oral health outreach importance. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest score and 10 being the highest. Higher score means better outcome. Then, we will average these composite scores for each group.
Attitudes Posttest Score | Posttest (2 weeks after baseline)
  We will ask all participants Likert-type scale questions about attitudes towards conducting oral health outreach. Each answer choice rating will range from 1 to 10, with higher ratings representing higher perceptions of oral health outreach importance. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest score and 10 being the highest. Higher score means better outcome. Then, we will average these composite scores for each group.
Self-efficacy Pretest Score | Baseline
  We will ask all participants Likert-type scale questions related to perceived self-efficacy with conducting oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceptions of confidence in providing oral health outreach. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, we will average these composite scores for both groups.
Self-efficacy Posttest Score | Posttest (2 weeks after baseline)
  We will ask all participants Likert-type scale questions related to perceived self-efficacy with conducting oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceptions of confidence in providing oral health outreach. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, we will average these composite scores for both groups.
Intentions Pretest Score | Baseline
  We will ask all participants Likert-type scale questions related to their intentions to conduct oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceived likelihood of providing oral health outreach in the future. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, we will average these composite scores for each group.
Intentions Posttest Score | Posttest (2 weeks after baseline)
  We will ask all participants Likert-type scale questions related to their intentions to conduct oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceived likelihood of providing oral health outreach in the future. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, we will average these composite scores for each group.
Skills Pretest Score | Baseline
  We will ask all participants Likert-type scale questions related to their skills to conduct oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceived skills to providing oral health outreach in the future. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, we will average these composite scores for each group
Skills Posttest Score | Posttest (2 weeks after baseline)
  We will ask all participants Likert-type scale questions related to their skills to conduct oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceived skills to providing oral health outreach in the future. We will average ratings from each question to create an average composite rating for each participant ranging from 0 to 10, with 0 being the lowest possible score and 10 being the highest score. Higher scores mean better outcomes. Then, we will average these composite scores for each group

SECONDARY OUTCOMES:
Satisfaction at posttest score | Posttest (2 weeks after baseline)
  We will ask only the intervention group participants Likert-type scale questions related to their satisfaction with the GRIN course. Each rating will range from 1 to 10, with higher scores representing higher satisfaction with the GRIN intervention. We will average ratings from each question to create an average composite rating for each intervention participant, then we will average these scores across the intervention group. Scores ranged from 1 to 10, with higher scores meaning better satisfaction/outcome.

OTHER OUTCOMES:
Change in Knowledge Scores From Pretest to Posttest | From baseline to posttest (2 weeks)
  At both pretest and posttest, we will ask all participants the same multiple choice knowledge questions related to oral health, which we will average to create a composite knowledge score for each participant ranging from 0 to 100. A score of 0 means a participant got zero questions correct while a score of 100 means a participant got all questions correct. We will average these composite scores across all participants for both groups to create mean scores. We will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Attitude Scores From Pretest to Posttest | From baseline to posttest (2 weeks)
  At both pretest and posttest, we will ask all participants Likert-type scale questions about attitudes towards conducting oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceptions of oral health outreach importance. We will average ratings from each question to create an average composite rating for each participant, then average these composite scores for both groups. We will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Self-efficacy Scores From Pretest to Posttest | From baseline to posttest (2 weeks)
  At both pretest and posttest, we will ask all participants Likert-type scale questions related to perceived self-efficacy with conducting oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceptions of confidence in providing oral health outreach. We will average ratings from each question to create an average composite rating for each participant, then average these composite scores for both groups. We will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Intentions Scores From Pretest to Posttest | From baseline to posttest (2 weeks)
  We will ask all participants Likert-type scale questions related to their intentions to conduct oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceived likelihood of providing oral health outreach in the future. We will average ratings from each question to create an average composite rating for each participant, then average these composite scores for both groups. We will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.
Change in Skills Scores From Pretest to Posttest | From baseline to posttest (2 weeks)
  We will ask all participants Likert-type scale questions related to their skills to conduct oral health outreach. Each rating will range from 1 to 10, with higher ratings representing higher perceived likelihood of providing oral health outreach in the future. We will average ratings from each question to create an average composite rating for each participant, then averaged these composite scores for both groups. We will then subtract pretest scores from posttest scores and average these changes for all participants. Higher scores mean higher gains from baseline to posttest.

CONTACTS AND LOCATIONS:
Overall Officials: Dexter L Cooper, Principal Investigator — KDH Research & Communication
Locations (1):
- KDH Research & Communication, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT07147244/Prot_SAP_000.pdf